CLINICAL TRIAL: NCT05431192
Title: Targeting Cognitive Function and Interoceptive Awareness to Improve Self-management in Patients With Co-morbid Heart Failure and Cognitive Impairment.
Brief Title: Mind Your Heart-II
Acronym: MYH-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Senior Research Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R01AG076438 (NIH); R01AG076438 (NIH)
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Cognitive Impairment
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be masked to intervention allocation. The PI, the co-investigators, and personnel responsible for data management and analysis will be blinded to participants' exposure status.
  Unblinded personnel will include the PD, the RA, and the MT instructors. Blinding the PD would be impossible given that she will be responsible for randomization and AEs monitoring.
  The RA will be responsible for data collection and will not be blinded. We note, however, that study participants will independently perform all assessments via computer interface with no RA involvement.
  The mindfulness instructors will be aware of the allocation status of the participants but will remain masked to the study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Training + Enhanced Usual Care (Experimental): Participants will receive a 30-minute, individual, phone-delivered session once a week for 8 weeks.
  Interventions: Behavioral: Mindfulness Training + Enhanced Usual Care
- Enhanced Usual Care alone (Other): Usual care.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Mindfulness Training + Enhanced Usual Care — Participants will receive a 30-minute, individual, phone-delivered session once a week for 8 weeks. MT involves training in the following (1) Awareness of breath; (2) Body scan; (3) Directing attention to simple activities of daily life; (4) Becoming aware of own thoughts and emotions; (5) "Open awareness" - a technique by which the participant is invited to direct his/her attention to any event arising in their field of experience at a given moment.
  In addition, participants will practice mindfulness techniques for 20 minutes daily on their own with the guidance of a digitally recorded, standardized guided mindfulness practice.
  Arms: Mindful Training + Enhanced Usual Care
Other: Enhanced Usual Care — Usual care will be enhanced in BOTH conditions with printed education materials provided to all participants using publicly available materials (the "Healthier Living with Heart Failure" guide available at the AHA Heart Failure Resource Center).66 The guide is organized in 7 chapters containing information on topics such as understanding HF, making healthy lifestyle changes, managing HF symptoms, taking medications, and living well with HF. Printed materials will be mailed weekly to all participants during the first 8 weeks of the study.
  Arms: Enhanced Usual Care alone

SUMMARY:
This projects studies the role of mindfulness training (MT) to improve self-care among patients with heart failure and cognitive impairment.

DETAILED DESCRIPTION:
Stable outpatients patients with co-morbid heart failure (HF) and mild cognitive impairment (MCI) (n=176) will be randomly assigned to phone-delivered MT (a weekly, 30-minute session for 8 weeks integrated with 20-min daily guided individual practice via digital recordings) plus enhanced usual care (EUC) or to EUC alone. Per current recommendations, usual care will be enhanced in both groups with self-care education materials. At baseline, 3 months (end of treatment), and 9 months since baseline participants will undergo comprehensive assessments of cognitive function, psycho-behavioral factors, cardiac vagal control, and HF biomarkers.

This study has the following objectives:

1. To study the role of MT in improving cognitive function and HF self-care in patients with co-morbid HF and MCI. We hypothesize: 1a) Cognitive function will improve in MT vs. EUC at end of treatment (3 months); 1b) Improvements in cognitive function at end of treatment will mediate effects on self-care and HF biomarkers at follow-up (9 months since baseline).
2. To study the role of MT in improving interoceptive awareness and HF self-care in patients with co-morbid HF and MCI. We hypothesize: 2a) Interoceptive awareness will improve in MT vs. EUC at 3 months, and 2b) Changes in interoceptive awareness at end of treatment will mediate improvements in self-care and HF biomarkers at 9 months follow-up.
3. To study the mechanistic pathway linking MT, vagal control and cognitive function. We hypothesize: 3a) Vagal control will improve in MT vs. EUC at end of treatment (3 months); 3b) Changes in vagal control will mediate improvements in cognitive performance at 9 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* A documented diagnosis of HF
* Access to a telephone
* Mild cognitive impairment (MoCA score < = 26)
* Ability to understand and speak English or Spanish

Exclusion Criteria:

* Unwillingness/inability to provide informed consent
* Reversible causes of HF (e.g., takotsubo syndrome; myocarditis)
* Severe hearing impairment not allowing phone delivery
* Suicidal ideation or plan
* Current (at least once a month) mind/body practice
* Planning to move out of the area during the study period
* Severe cognitive impairment (MoCA scores < 15)
* New York Heart Association (NYHA) class IV heart failure or clinically unstable
* Ongoing psychiatric or neurologic conditions
* Current enrollment in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in average Fluid Cognition Composite score from the NIH Toolbox Fluid Cognition Battery. | Baseline, 3 months, 9 months
  The NIH Toolbox is comprised of seven cognitive tests, of which two measure crystallized cognitive ability (i.e., vocabulary and reading) and five tests measure fluid cognitive functioning (i.e., working memory, memory, speed of processing, and executive function). The fluid cognition composite score is obtained by averaging the normalized scores of the Fluid Cognition measures. Higher scores indicate higher levels of functioning. A score ~ 100 indicates average fluid cognitive ability compared with others nationally. Scores ~115 suggest above-average ability, while scores ~130 suggest superior ability. Conversely, a score in the range of 85 suggests below-average ability, and a score ~ 70 or below suggests significant impairment.

SECONDARY OUTCOMES:
Change in average Multidimensional Assessment of Interoceptive Awareness (MAIA) scores. | Baseline, 3 months, 9 months
  The MAIA is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. Higher scores on each subscale indicate higher levels of interoceptive awareness.There are no standard normal values for each MAIA sub-scale; the range in previous samples from our group for the Not Distracting Score was 1-14. ; MAIA: Not Worrying Score 4-13; MAIA: Attention Regulation Score 4-35; MAIA: Emotional Awareness Score 5-25; MAIA: Self-Regulation Score 4-20; MAIA: Body Listening Score 1-15; MAIA: Trusting Score 3-15.
Change in average Heart Failure (HF) Self-Care total scores. | Baseline, 3 months, 9 months
  The Self-care of HF Index (SCHFI) v.7.2., is a psychometrically valid, self-report instrument with three separate scales: Self-Care Maintenance (which captures treatment adherence and healthy behaviors), Symptom Perception (which assesses the ability to detect and interpret physical symptoms), and Self-Care Management (the response to symptoms when they occur). Reliability is > 0.70 and scores range from 0 to 100; higher scores indicate better self-care.
Change in average Depression subscale score on the Hospital Anxiety and Depression Scale (HADS). | Baseline, 3 months, 9 months
  The HADS is a self-reported measure with two sub-scales (scores 0-21) measuring anxiety and depression, with higher scores indicating greater psychological morbidity. A good correlation has been reported between the HADS and other commonly used measures of depression. The HADS has been validated in cardiac patients.
Change in average Kansas City Cardiomyopathy Questionnaire (KCCQ) Health Scores. | Baseline, 3 months, 9 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) quantifies HF-specific physical limitations, symptom frequency, severity and change over time, overall quality of life, social interference, and knowledge. Responses are scored on a Likert scale and summed. Higher scores indicate higher quality of life. Construct validity and sensitivity of the KCCQ have been demonstrated.
Change in high frequency power heart rate variability (hf-HRV) in Ln msec2. | Baseline, 3 months, 9 months
  High-frequency band is an index of cardiovagal control. High frequency power (hf-HRV) in Ln msec2 , a demonstrated index of vagal activity, will be determined by averaging high frequency values for 10 minute segments at each visit. The proposed methods are based on standards established in the literature.
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP)levels. | Baseline, 3 months, 9 months
  NT-proBNP is a marker of HF disease severity, elevated filling pressures, clinical outcomes, and is responsive to interventions (e.g., exercise). Specimens are collected in a plastic EDTA tube , centrifuged and separated plasma samples are stored at -20°C until testing. Assays will be analyzed using the ADVIA Centaur BNP assay, a fully automated two-site sandwich immunoassay using direct chemiluminescent technology . The ADVIA Centaur BNP assay measures BNP concentrations up to 5000 pg/mL with a minimum detectable concentration (analytical sensitivity) of < 2.0 pg/mL and shows high specificity for BNP.
Change in average 6-min walk test (6MWT) distance. | Baseline, 3 months, 9 months
  The 6MWT measures the distance a patient can walk on a level course in 6 min. It is a measure of functional capacity that correlates with peak oxygen uptake and is positively associated with survival in patients with cardiovascular disease. A higher value (in meters) indicates better functional capacity. The 6MWT distance in healthy adults has been reported to range from 400 to 700 meters.

OTHER OUTCOMES:
HF hospital readmissions | 9 months
  Proportion of patients admitted to the hospital with a diagnosis of HF. HF hospital admissions will be tracked via EMR and direct inquiry with participants.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, MD, PhD, Principal Investigator — Cardiovascular Institute, The Miriam Hospital, Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under the project will be shared as per the NIH Grant Policy and The Miriam Hospital IRB guidelines. Deidentified research data will be made available in a timely manner once the main findings from the final research data set have been accepted for publication. Access to these data will be available for educational or research purposes. Data will be deidentified to avoid linkages to individual research participants and will not contain variables that could lead to the disclosure of the identity of individual subjects. All requestors will be asked to sign a data sharing agreement that includes conditions to 1) protect the identity of participants, 2) limit use of data for educational and research purposes, 3) prevent transfer of data to other users, and 4) acknowledge the data source. The de-identified data will be shared using Excel or SPSS file formats.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once the main findings from the final research data set have been accepted for publication.
Access Criteria: Researchers interested in obtaining the de-identified data and associated documentation (e.g. analytical code) can make a request to the principal investigator by email.